CLINICAL TRIAL: NCT05171036
Title: Etude Des éléments Posturographiques Statiques et Dynamiques prédictifs de la Chute de la Personne âgée institutionnalisée
Brief Title: Study of Static and Dynamic Posturographic Elements Predictive of Falls in the Institutionalized Elderly
Acronym: POSTADYCHUTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Borelli UMR 9010 (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ID-RCB 2017-A02545-48
Record Dates: First submitted 2021-11-25; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Fall; Aging; Gait, Unsteady; Motor Activity
MeSH Terms: conditions — Gait Disorders, Neurologic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Institutionalized elderly people undergoing adapted physical activity (Experimental): 2h/week for 3 months (i.e. 24 sessions), after 3 months of no-APA for gait and balance baseline recordings, with the rehabilitation team in place in the establishments, around the 4 specific programmes
  Interventions: Other: Adapted Physical Activity

INTERVENTIONS:
Other: Adapted Physical Activity — * Group 1 Maintenance of autonomy: "Patients in group 1 have no cardiovascular disorders, possibly some cognitive deficits but do not reside in a protected unit.
  * Group 2 Prevention of the risk of falls: "Patients in group 2 have no cardiovascular problems, possibly some cognitive problems, but can finally follow the indications of the cognitive assessment in the form developped for the study.
  * Group 3 Prevention of the risk of falls and monitoring of cardiovascular disorders in the absence of cognitive impairment: "Patients in group 3 have had a recent, and currently stabilised, cardiovascular event that may justify exercise reconditioning.
  * Group 4 Prevention of the risk of falls and disorientation in a context of cognitive deficit: "Patients in group 4 have moderate to severe cognitive disorders, or have Alzheimer's disease or a related disease at a stage of the disease requiring special attention.

SUMMARY:
A fall in the elderly is defined by the WHO as "an event in which a person [over 65 years of age] inadvertently falls to a lower level on the ground or other surface than they were previously at". The severity of the consequences of falls is correlated with the age of the person who suffers them, making people over 65 at risk. Since 2000, the number of falls among the elderly has not decreased, including in institutions. Today, the direct and indirect costs of falls are estimated at 1.7 billion euros in France.

The French National Authority for Health (HAS) stresses that the lack of success of prevention policies is due in particular to the lack of evaluation and prevention resources. In nursing homes, this lack of resources is sometimes used to justify passive restraint to ensure the safety of participants. However, this method poses the problem of the free movement of residents within the institution. The fall detection technologies already on the market do not allow for the assessment of the risk of falling and therefore for early action.

Based on the latest scientific data in static posturography, researchers at the Borelli Centre have developed posturographic markers whose non-linear analysis makes it possible to establish an objective and clinically relevant score based on the study of the displacement of the centre of pressure. In contrast to the techniques commonly used in the laboratory to study balance (which are not usable in health care institutions because of their cost, lack of transportability and the expertise required to explore the recorded data), this method of measurement allows health care professionals to quickly and easily measure the balance of participants in routine consultations. Thus, special attention and targeted rehabilitation can then be implemented to prevent falls and their consequences.

DETAILED DESCRIPTION:
Since 2000, the number of falls among the elderly has not decreased, even in institutions. The HAS stresses that the lack of success of prevention policies is due in particular to the lack of means of evaluation and prevention. Based on the latest scientific data in static posturography, researchers at the UMRD Cognac-G have developed posturographic markers whose non-linear analysis makes it possible to establish an objective and clinically relevant score for analysing the risk of falls in EHPAD residents. This measurement method, patented [FR1660846; FR1660850; FR1557582; FR1770031] and published [Oudre, 2015; Audiffren, 2016; Barrois, 2017; Bargiotas, 2018], allows health professionals to quickly assess the balance of participants in routine consultations.

According to the WHO, falls are the consequence of many multidimensional factors. Adapted physical activity can have a beneficial effect on these factors, particularly in terms of reducing risk behaviours, modifying the environment and improving physiological capacities. If the results of the study prove to be relevant, in the long term, measurements based on the Borelli Centre's method of measuring balance in EHPAD could be recommended. It could thus help doctors in the early management of balance disorders in institutionalized elderly people.

The main objective of this Postadychute-AG study is to quantify and monitor the risk of falls in the elderly on a monthly basis by validating the relevance of the patented indicators and their analysis, which are obtained from a statokinesigram recorded on a force platform and data from inertial units measuring the movements of body segments, predicting the risk of falling. This will be done by comparing the predicted risk of falling with the number of falls actually recorded each month of follow-up of institutionalized seniors undergoing adapted physical activity (APA). Our secondary objectives are also to :

* To study the sensitivity of our model to the natural evolution of nursing home residents during a 3-month observation period without APA and to the improvement of their condition with APA sessions in addition to routine care
* To assess the acceptability of the measurement method and the use of the fall score through the scale developed for this purpose among nursing home staff.
* If the results of the study prove to be relevant, the ultimate aim is to recommend that measurements be taken using the measurement method used in this study. It will thus be able to help doctors in their diagnosis and early management of balance disorders by teams of rehabilitation specialists.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects of both sexes, aged 65 and over, with social insurance;
* Residing in an ORPEA Group retirement home;
* Do not have a neurological, inner ear or visual disorder that is incompatible with climbing on the force platform or walking 10 metres round trip without human assistance;
* Can safely climb onto the platform by force (as estimated by the investigating practitioner) and can maintain an erect position for more than 1 minute, with eyes open or closed;
* Had an MMSE score of more than 18 on the nursing home entrance examination;
* Having a life expectancy of more than 6 months, as estimated by the coordinating doctor;
* Having signed the informed consent.

Non-inclusion Criteria:

* Non-mobile resident: any person with a musculoskeletal or neurosensory disorder that does not allow them to stand for more than 1 minute on the power platform;
* History of limb amputation;
* Blindness, assessed using an Amsler grid;
* Refusal of the resident.

Exclusion Criteria:

* Exit from the trial by resident's choice ;
* Inability of the resident to continue with static and dynamic assessments (e.g. due to a serious adverse event following a fall) The study is an intention-to-treat study and data from participants who do not complete the protocol will be used until the date of their exclusion from the trial or their death.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2022-01-17 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of indicators measured monthly over the 6 months of follow-up | Every 6 months
  Predictive value of indicators measured monthly over the 6 months of follow-up (3 months without ABS followed by 3 months with ABS). The predictive value will be quantified by an evaluation of the threshold of the predictive score out of 100, based on a minimum sensitivity of 80% and a maximum specificity (the Youden index is the numerical criterion), via an ROC curve and a measurement of the area under the curve (AUC) for the classification between "at high risk of falling" and "at low risk of falling" (binary criterion). This classification is subsequently verified by means of the falls collection sheets and the falls history at the next visit.

SECONDARY OUTCOMES:
Positive (PPV) and Negative (NPV) predictive values based on the binary classification "high risk of falling" and "low risk of falling". | Every 6 months
  As with the AUC, PPV and NPV will be calculated on the basis of the questionnaires and the falls form recorded each month. This method has been used previously to assess the predictive qualities of clinical tests.
Correlation of fall risk indicators with other recorded variables | Every 6 months
  A value of more than 0.7 and a significance of the correlation test will be considered as indicating a strong correlation between the predictive score on the one hand and falls in the institution or the clinical course of the participants on the other.

OTHER OUTCOMES:
Acceptability of the measure system | At 24 months
  The acceptability of the use of the predictive score will be measured via the predictive score form at the end of the 6-month follow-up. This questionnaire is based on the Technology Acceptance Model and the 7-point Likert scale. The questionnaire will be sent to the rehabilitation teams and the coordinating doctors of the institutions. A high score represents a high degree of aggreement. Each of the 24 items is scored from 1 to 7, with 1 representing a "total disagreement" with the statement and 7 a "total agreement". The score ranges from 24 to 168 points.

CONTACTS AND LOCATIONS:
Overall Officials: Flavien QUIJOUX, PhD, Principal Investigator — Orpea Group

IPD SHARING:
Plan to Share IPD: Yes
The clinical trial data will be aggregated and presented as averages by group and subgroup in order to comply with the regulatory authorities in the treatment of so-called sensitive data, particularly in relation to the health and identity of the persons involved in the research.
  Scientific publications concerning the protocols, methods of analysis of the data used and the results of the study will be submitted to peer-reviewed journals and/or code-sharing platforms to promote reproducible and transparent science.
Supporting Information: Study Protocol, Analytic Code
Time Frame: 2021 - Publication of the Protocole 2022 - Publication of the preliminary results 2023/24 - Publication of the final results

REFERENCES:
- [Background] Quijoux F, Bertin-Hugault F, Zawieja P, Lefevre M, Vidal PP, Ricard D. Postadychute-AG, Detection, and Prevention of the Risk of Falling Among Elderly People in Nursing Homes: Protocol of a Multicentre and Prospective Intervention Study. Front Digit Health. 2021 Jan 27;2:604552. doi: 10.3389/fdgth.2020.604552. eCollection 2020. PMID 34713067
- [Background] Quijoux F, Vienne-Jumeau A, Bertin-Hugault F, Zawieja P, Lefevre M, Vidal PP, Ricard D. Center of pressure displacement characteristics differentiate fall risk in older people: A systematic review with meta-analysis. Ageing Res Rev. 2020 Sep;62:101117. doi: 10.1016/j.arr.2020.101117. Epub 2020 Jun 19. PMID 32565327
- [Background] Dot T, Quijoux F, Oudre L, Vienne-Jumeau A, Moreau A, Vidal PP, Ricard D. Non-Linear Template-Based Approach for the Study of Locomotion. Sensors (Basel). 2020 Mar 30;20(7):1939. doi: 10.3390/s20071939. PMID 32235667